CLINICAL TRIAL: NCT00464217
Title: PETHEMA-LAM99:Treatment of the Acute Myeloblastic Leukaemia in Patients Over 65 Years
Brief Title: Treatment of the Acute Myeloblastic Leukaemia in Patients Over 65 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETHEMA/LAM-99
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Acute Myeloblastic Leukaemia
Keywords: Acute Myeloblastic Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; molgramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ARA-C
Drug: Idarubicin
Drug: Leucomax

SUMMARY:
To reproduce or to improve the index of complete responses of protocol LMA-91 with a similar protocol, decreasing the dose of Idarubicin to try to reduce the deaths in induction

DETAILED DESCRIPTION:
INDUCTION TREATMENT :Ara-C 100 mg/m 2 /day in continuous perfusion,days 1 - 7. Idarubicin 8 mg/m 2 /day, days 1 - 3 in bolus. GM-CSF (Leucomax) 5 mcg/kg subcutaneous or endovenous from day + 4 after finishing the chemotherapy until the recovery of neutropenia (> 1.000/mm 3)

CONSOLIDATION TREATMENT The patients who reach a complete response with the first cycle, will receive a second cycle to consolidation. The patients who do not reach a complete response with the first cycle will receive a second cycle. If after two cycles,do not obtain the response, patient should leave the protocol.

INTENSIFICATION TREATMENT All the patients who are in complete response after one cycle of induction and one cycle of consolidation, or after two cycles of induction, will receive a treatment of intensification with: ARA-C 500 mg/m 2 /12 h in one hour infusion, days 1-4. Daunomycin 45 mg/m 2 /day bolu, days 5-7. GM-CSF (Leucomax): 5 mcg/kg from day to + 4 after finishing the chemotherapy until the recovery of neutropenia (>1.000/mm 3)

ELIGIBILITY:
Inclusion Criteria:

* Cytologic diagnosis of acute myeloblastic leukaemia (excluded M3)
* Over 65 years

Exclusion Criteria:

* Previous diagnosis of other malignancy hematopoietic disorder or myelodysplastic syndrome
* Previous treatment with antileucemic chemotherapy
* Psychiatric disorder
* Diagnosis of subtype FAB M3
* Creatinine > 2.5 mg/dL
* Bilirubin , Alkaline Phosphatase or transaminases three times upper the limit

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100
Dates: Start 1998-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Improve the complete response index in patients diagnosed of acute myeloblastic leukaemia over 65 years

SECONDARY OUTCOMES:
Evaluate the toxicity
Evaluate the effect of haematopoietic growth factors

CONTACTS AND LOCATIONS:
Overall Officials: Garcia Laraña Jose, Dr, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (24):
- Spain (24):
  - Hospital General de Albacete, Albacete
  - Hospital Universitario, Alicante
  - Hospital Puerta del Mar, Cadiz
  - Hospital Ntra. Sra. del Rossell, Cartagena
  - Hospital General, Castellon
  - Hospital de Galdacano, Galdakao
  - Hospital Ciudad de Jaén, Jaén
  - Hospital Insular de las Palmas, Las Palmas de Gran Canaria
  - Hospital Xeral, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario de Alcalá de Henares, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Messeguer, Murcia
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Central de Asturias, Oviedo
  - Clínica Universitaria de Pamplona, Pamplona
  - Hospital Montecelo, Pontevedra
  - Hospital Clínico Universitario, Salamanca
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínico, Valencia
  - Hospital Dr. Pesset, Valencia
  - Hospital Clínico, Valladolid
  - Hospital Virgen de la Concha, Zamora

REFERENCES:
- [Derived] Martinez-Lopez J, Fernandez-Redondo E, Garcia-Sanz R, Montalban MA, Martinez-Sanchez P, Pavia B, Mateos MV, Rosinol L, Martin M, Ayala R, Martinez R, Blanchard MJ, Alegre A, Besalduch J, Bargay J, Hernandez MT, Sarasquete ME, Sanchez-Godoy P, Fernandez M, Blade J, San Miguel JF, Lahuerta JJ; GEM (Grupo Espanol Multidisciplinar de Melanoma)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) cooperative study group. Clinical applicability and prognostic significance of molecular response assessed by fluorescent-PCR of immunoglobulin genes in multiple myeloma. Results from a GEM/PETHEMA study. Br J Haematol. 2013 Dec;163(5):581-9. doi: 10.1111/bjh.12576. Epub 2013 Oct 3. PMID 24117042
- See also: Spanish association of Haematology — http://www.aehh.org